CLINICAL TRIAL: NCT03261661
Title: Improving Response to Intervention in Students With or at Risk of Reading Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Southern Methodist University (Other); Florida State University (Other)
Responsible Party: Principal Investigator, Jeanne Wanzek, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170686
Record Dates: First submitted 2017-08-07; First posted 2017-08-25 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Reading Problem
MeSH Terms: interventions — Stress Mindset Measure; Commerce

STUDY DESIGN:
Intervention Model Description: Random assignment through stratification on the screening score to one of three groups: Study 1: (a) Reading Intervention Plus Mindset, (b) Reading Intervention, or (c) Business as Usual comparison.
  Study 2: (a) Reading Intervention Embedded with Mindset or (b) Business as Usual comparison.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Reading Plus Mindset (Experimental): Multicomponent reading intervention providing explicit and systematic instruction in phonological awareness, phonics and word recognition, and reading fluency. Participants also complete mindset training and activities.
  Interventions: Behavioral: Reading; Behavioral: Mindset
- Reading Embedded with Mindset (Experimental): Multicomponent reading intervention (providing explicit and systematic instruction in phonological awareness, phonics and word recognition, and reading fluency) with mindset instruction specific to reading progress embedded in the intervention Participants also complete mindset training and activities.
  Interventions: Behavioral: Reading; Behavioral: Mindset; Behavioral: Reading Embedded with Mindset
- Reading (Active Comparator): Multicomponent reading intervention providing explicit and systematic instruction in phonological awareness, phonics and word recognition, and reading fluency.
  Interventions: Behavioral: Reading
- Business as Usual (Active Comparator): Participation in the typical reading instruction and intervention provided within participating schools.
  Interventions: Behavioral: Business as Usual

INTERVENTIONS:
Behavioral: Reading — Students are taught the processes involved in hearing, seeing, and feeling sounds as well as differences between sounds in words. New knowledge is built on previous knowledge in a step-by-step manner. Sounds build to letter-sound relationships to reading of words and syllables. Students learn the connection between reading of words (decoding) and writing/spelling words (encoding) building from simple words to multisyllabic words to text reading with fluency and understanding.
  Arms: Reading; Reading Embedded with Mindset; Reading Plus Mindset
Behavioral: Mindset — Blended learning program with online and teacher-directed activities related to how the brain functions, learns, and remembers, and how it changes in a physical way when we exercise it. Instruction in how students are in control of their brain and its development, and how to apply this to their schoolwork with practical strategies for tackling academic challenges.
  Arms: Reading Embedded with Mindset; Reading Plus Mindset
Behavioral: Reading Embedded with Mindset — Mindset training explicitly linked to the reading content through lesson openers, feedback prompts, and self-monitoring of mindset during reading work.
  Arms: Reading Embedded with Mindset
Behavioral: Business as Usual — Reading interventions already provided to students with reading difficulties as per typical procedures at the participating school
  Other Names: Typical Instruction
  Arms: Business as Usual

SUMMARY:
The purpose of the proposed studies is to examine a reading intervention for fourth grade students with reading difficulties that integrate work in mindset (beliefs about whether abilities are innate or can be developed) with the academic component of reading. Specifically, the investigators will examine the extent to which integrating mindset intervention improves student response to reading intervention. The investigators will use previous research in intensive reading intervention for students with reading difficulties in the upper elementary grades to examine an intervention that addresses reading skill deficits, while also providing mindset training along with (Study 1) or embedded in (Study 2) the reading intervention. It is hypothesized that students in the reading intervention with mindset conditions will improve their reading outcomes more than students in the reading intervention only and business as usual groups.

DETAILED DESCRIPTION:
The purpose of the proposed studies is to examine a reading intervention for fourth grade students with RD that integrates the psychosocial component of mindset with the academic component of reading. Specifically, the investigators will examine the extent to which integrating mindset intervention improves student response to reading intervention. The investigators will use previous research in intensive reading intervention for students with RD in the upper elementary grades to examine an intervention that addresses reading skill deficits, while providing mindset training along with (Study 1) or embedded in (Study 2) the reading intervention.

Specific Aim 1. To determine the effects of intensive reading intervention with mindset training (Reading Intervention Plus Mindset) relative to reading intervention alone and business as usual comparison on the academic outcomes of fourth grade students with or at-risk for reading disabilities. The proposed study will target students with or at-risk for reading disabilities in fourth grade to examine the effects of reading intervention with mindset training relative to reading intervention alone and business as usual comparison on students' mindset, general academic achievement, phonological awareness, word reading, fluency, and reading comprehension outcomes. Students will be randomly assigned to condition with students in the Reading Intervention Plus Mindset condition receiving the mindset training along with their reading intervention. Students assigned to the Reading Intervention will receive the same reading intervention but without the mindset training. Students in the Business as Usual condition will continue to receive their typical school services which will be carefully documented. It is hypothesized that students in the Reading Intervention Plus Mindset condition will improve their reading outcomes more than students in the Reading Intervention only and Business as Usual groups by continuing to develop a growth mindset to work through the challenges in their reading development and, thus, being able to progress more efficiently in the reading intervention.

Specific Aim 2. To determine the effects of embedding mindset training in an intensive reading intervention on the mindset and academic outcomes of fourth grade students with or at-risk for reading disabilities. The proposed study will use the results from Specific Aim 1 to further examine the effects of an intensive reading intervention with mindset embedded in the content with a new cohort of fourth grade students with or at-risk for reading disabilities. Embedding mindset practices directly in the content area of difficulty for students with learning difficulties could be more powerful than separate mindset training. Students will be randomly assigned to one of two conditions (Embedded or Business as Usual). The investigators will examine the effects of intervention on students' mindset, word reading, fluency, and reading comprehension measures. It is hypothesized that embedding mindset training directly in the reading content will further improve student reading outcomes by allowing students to directly apply a growth mindset to their work in the area of difficulty, reading.

Specific Aim 3. To link student characteristics to response to intervention. The proposed study will link students' initial reading achievement, initial mindset, vocabulary ability, behavior/attention as well as race, sex, socioeconomic status, and parents' educational background to student response to intervention. It is hypothesized that students with lower initial reading achievement, higher initial levels of fixed mindset, higher vocabulary, lower parent educational background or socioeconomic status, and/or higher levels of problem behavior/attention initially will benefit more from the mindset intervention, particularly the embedded mindset intervention. It is hypothesized that no differences based on gender or race.

ELIGIBILITY:
Inclusion Criteria:

Fourth grader Identified with reading difficulty

-

Exclusion Criteria:

Identified vision, hearing, or intellectual disability

-

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 580 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Cloze Reading Comprehension | baseline, within 3 weeks of intervention completion
  Students are instructed to read a short passage and identify a missing key word that would make sense
Change in Passage Reading Comprehension Study 1 only | baseline, within 3 weeks of intervention completion
  The comprehension assessment consists of expository and narrative passages that increase in length, followed by multiple choice questions.
Change in Word Reading | baseline, within 3 weeks of intervention completion
  Students reads a list of real words
Change in Decoding | baseline, within 3 weeks of intervention completion
  Student reads a list of nonsense words
Change in Reading Fluency | baseline, within 3 weeks of intervention completion
  Students read three passages aloud for 1 min. The total number of correct words is counted.
Change in Phonological Processing Blending Study 1 only | baseline, within 3 weeks of intervention completion
  Blending requires the students to listen to a series of real words spoken in segments and earn a point for each word they blend correctly.
Change in Phonological Processing Deletion Study 1 only | baseline, within 3 weeks of intervention completion
  Elision requires a student to listen to a segmented word and then pronounce the word without a segment.
Change in Word Reading Fluency | baseline, within 3 weeks of intervention completion
  Students reads a list of real words. The number of words read in 45 seconds is counted
Change in Decoding Fluency | baseline, within 3 weeks of intervention completion
  Student reads a list of nonsense words. The number of words read in 45 seconds is counted

SECONDARY OUTCOMES:
Mindset | baseline, within 3 weeks of intervention completion
  Ratings of how student thinks about learning and the brain
Change in Math Problem Solving Study 1 only | baseline, within 3 weeks of intervention completion
  Students analyze and solve math problems

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Vanderbilt University, Nashville, Tennessee
  - Southern Methodist University, Dallas, Texas